CLINICAL TRIAL: NCT05408780
Title: A Phase 1, Two-part, Randomized Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Liquid Formulation of Tricaprilin, and Matching Placebo to Include Single-dose and Food Effect (Part A), and Titration Tolerability (Part B), in Healthy Subjects
Brief Title: A Phase 1, Two-part, Randomized Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of a Liquid Formulation of Tricaprilin and Matching Placebo in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: AC-22-028
Record Dates: First submitted 2022-05-31; First posted 2022-06-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This is a two-part study.
  Part A (Food Effect Assessment): It is a randomized, double-blind (to IMP received), placebo-controlled, four-period, single-dose design. Subjects will be dosed in the fed state or the fasted state depending on the regimen.
  Part B (Titration Tolerability): Participants will be administered to either tricaprilin or a matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A - Food Effect Assessment (Experimental): Subjects will be randomized before administration of the first dose of active or matching placebo IMP in a 1:1:1:1 ratio to 1 of 4 treatment sequences (ABCD, BACD, ABDC, BADC) so that all subjects receive Regimens A, B, C and D across the 4 periods.
  Interventions: Drug: AC-OLE-01-VA
- Part B - Titration Tolerability (Experimental): Subjects will be dosed BID in the morning and afternoon (approximately 5 h apart) on Days 1 to 27. Both doses of active or matching placebo IMP will be administered in the fed state either 30 min after completion of a standard-fat and calorie content breakfast or 30 min after a standardized-fat and calorie content lunch.
  Participants will be randomised to either study drug or the matching placebo.
  Interventions: Drug: AC-OLE-01-VA

INTERVENTIONS:
Drug: AC-OLE-01-VA — formulation of tricaprilin or matching placebo

SUMMARY:
The purpose of this study is to evaluate the PK, safety, and tolerability of a new liquid formulation of tricaprilin.

ELIGIBILITY:
Main Inclusion Criteria:

* Healthy males and non-pregnant, non-lactating healthy females aged 18 to 55 years inclusive at time of signing informed consent with a body weight ≥55 kg.
* Body mass index (BMI) 18.0 to 32.0 kg/m2 as measured at screening or, if outside the range, considered not clinically significant by the investigator.

Main Exclusion Criteria:

* Serious adverse reaction or serious hypersensitivity to any drug or formulation excipients
* Subjects with a history of fainting, dizziness, bradycardia or hypotension as considered clinically significant by the investigator
* Subject has a medical condition that may adversely affect taste or smell activity

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-08-13 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) of total ketones (β-hydroxybutyrate and acetoacetate) after single-dose administration of tricaprilin and placebo formulations (Part A) | 0 to 8 hours post-dose
  AUC will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)
Incidence of Treatment Emergent Adverse Events (Part B) | Baseline to 28 days
  Adverse event incidence will be tabulated

SECONDARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (Part A) | Baseline to 8 days
  Adverse event incidence will be tabulated [BARF] Scale)
Area under the concentration-time curve (AUC) of total ketones (β-hydroxybutyrate and acetoacetate) of tricaprilin and placebo formulations following a titration scheme (Part B) | 0 to 8 hours post-dose
  AUC will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)
Maximum observed concentration (Cmax) of total ketones (β-hydroxybutyrate and acetoacetate) after administration of tricaprilin and placebo formulations (Part A, Part B) | 0 to 8 hours post-dose
  Cmax will be calculated from PK concentrations of total ketones (B-hydroxybutyrate and Acetoacetate)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Cerecin
Locations (1):
- Quotient Sciences Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No